CLINICAL TRIAL: NCT04508062
Title: Effects of the Addition of Uterosacral Ligament Plication to Pectopexy Operation on Anatomical and Subjective Symptoms in the Treatment of Apical Compartment Defects
Brief Title: Effects of the Addition of Uterosacral Ligament Plication to Pectopexy Operation on Anatomical and Subjective Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Gamze Nur Cimilli Şenocak, assistant professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B.30.2.ATA.0.01.00/6
Record Dates: First submitted 2020-05-29; First posted 2020-08-11 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Pelvic Organ Prolapse
Keywords: pelvic organ prolapse; pectopexy; laparoscopy; uterosacral ligaments plication
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pectopexy group (Active Comparator): this group will only have pectopexy operation
  Interventions: Procedure: pectopexy operation
- Pectopexy and uterosacral ligaments plication group (Active Comparator): this group will have pectopexy operation with bilateral uterosacral ligaments plication
  Interventions: Procedure: pectopexy operation; Procedure: uterosacral ligaments plication operation.

INTERVENTIONS:
Procedure: pectopexy operation — Vaginal cuff or uterine cervix will be attached to iliopectineal ligament with polypropylene mesh on both sides.
Procedure: uterosacral ligaments plication operation. — At least 2/3 of the sacrouterine ligaments will be shortened with helical sutures, starting from the cervix and so douglas will be partially obliterated.
  Arms: Pectopexy and uterosacral ligaments plication group

SUMMARY:
The investigators planned to measure the effectiveness of laparoscopic pectopexy in apical prolapse and whether the addition of sacrouterine ligaments plication to pectopexy increases the effectiveness of pectopexy operation. Investigators planned to measure patients' quality of life using the female sexual function scale test 3, 6 and 12 months after the surgery and to determine how the operation affects the quality of sexual life.

DETAILED DESCRIPTION:
In this study, the investigators planned to measure the effectiveness of laparoscopic pectopexy in apical prolapse and whether the addition of sacrouterine ligaments plication to pectopexy increases the effectiveness of pectopexy operation. Investigators planned to measure patients' quality of life using the female sexual function scale test 3, 6 and 12 months after the surgery and to determine how the operation affects the quality of sexual life.

ELIGIBILITY:
Inclusion Criteria:

* patients with stage II-IV apical compartment defect according to the POP-Q classification

Exclusion Criteria:

* having severe chronic disease that makes the operation dangerous
* patients under 25 and patients over 75 years old

Ages: 25 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2021-03-06 (Actual); Study Completion 2022-03-06 (Actual)

PRIMARY OUTCOMES:
questionnaire of lower urinary tract symptoms | changes in symptoms for each title at the preoperative day 1 and postoperative day 3 period
  the questionaire examines these titles by scoring from one to ten points:
  1. sudden feeling of ürination
  2. sudden feeling of urination with incontinence
  3. Frequent urination
  4. Difficulty of starting the urination
  5. Abnormal discharge of urine
  6. nocturia
  7. dyspareunia
  8. Stress urinary incontinence
  9. dysuria
  10. constipation
evaluation of sexual function with Women's Sexual Function Index | changes at the preoperative day 1 and postoperative day 40 period
  Women's Sexual Function Index is a questionnaire about sexual functions of the women. the index definex sexual functions with some questions and scorings.
Stage of apical compartment defect according to the Pelvic Organ Prolapse (POP-Q) classification | changes in the stage of apical compartment defect at the preoperative day 1 and postoperative day 3 period according to POP-Q clasification
  Stage of apical compartment defect according to the Pelvic Organ Prolapse (POP-Q) classification

SECONDARY OUTCOMES:
evaluation of sexual function with Women's Sexual Function Index | changes at 3,6 and 12. month after surgery
  Women's Sexual Function Index is a questionnaire about sexual functions of the women. the index definex sexual functions with some questions and scorings.
Stage of apical compartment defect according to the Pelvic Organ Prolapse (POP-Q) classification | changes at 3,6 and 12. month after surgery
  Stage of apical compartment defect according to the Pelvic Organ Prolapse (POP-Q) classification
questionnaire of lower urinary tract symptoms | changes in symptoms for each title at 3,6 and 12. month after surgery
  the questionaire examines these titles by scoring from one to ten points:
  1. sudden feeling of ürination
  2. sudden feeling of urination with incontinence
  3. Frequent urination
  4. Difficulty of starting the urination
  5. Abnormal discharge of urine
  6. nocturia
  7. dyspareunia
  8. Stress urinary incontinence
  9. dysuria
  10. constipation

CONTACTS AND LOCATIONS:
Overall Officials: Gamze Nur Cimilli Senocak, Principal Investigator — Ataturk University
Locations (1):
- Gamze Nur Cimilli Senocak, Erzurum, Turkey (Türkiye)